CLINICAL TRIAL: NCT01204294
Title: An Open Label, Randomised, Parallel Group Safety and Efficacy Study of Linagliptin (5 mg Administered Orally Once Daily) Over 52 Weeks in Patients With Type 2 Diabetes Mellitus and Insufficient Glycaemic Control Despite Background Mono-therapy With an Approved Antidiabetic Drug
Brief Title: Comprehensive Add on Study in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1218.78
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Results first posted 2013-01-23 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; Metformin

ARMS (7):
- Bigu+Lina (Experimental): biguanide plus linagliptin
  Interventions: Drug: Linagliptin
- Glin+Lina (Experimental): glinide plus linagliptin
  Interventions: Drug: Linagliptin
- Glit+Lina (Experimental): glitazone plus linagliptin
  Interventions: Drug: Linagliptin
- SU+Lina (Experimental): sulfonylurea plus linagliptin
  Interventions: Drug: Linagliptin
- A-GI+Lina (Experimental): alpha-glucosidase inhibitor plus linagliptin
  Interventions: Drug: Linagliptin
- SU+Met (Active Comparator): sulfonylurea plus metformin
  Interventions: Drug: Metformin
- A-GI+Met (Active Comparator): alpha-glucosidase inhibitor plus metformin
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Linagliptin — Linagliptin once daily
  Arms: Glin+Lina
Drug: Linagliptin — Linagliptin once daily
  Arms: Glit+Lina
Drug: Metformin — Metformin twice or three time per day
  Arms: A-GI+Met
Drug: Metformin — Metformin twice or three time per day
  Arms: SU+Met
Drug: Linagliptin — Linagliptin once daily
  Arms: A-GI+Lina
Drug: Linagliptin — Linagliptin once daily
  Arms: Bigu+Lina
Drug: Linagliptin — Linagliptin once daily
  Arms: SU+Lina

SUMMARY:
The objective of the current study is to investigate the safety and efficacy of linagliptin (5mg / once daily) given for 52 weeks as add-on therapy to patients with type 2 diabetes mellitus and insufficient glycaemic control despite diet, exercise, and treatment with one approved antidiabetic drug.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of type 2 diabetes mellitus
2. Male and female patients on diet and exercise regimen who are treated with one antidiabetic drug

Exclusion criteria:

1. Myocardial infarction, stroke, transient ischemic attack, or pulmonary embolism
2. Impaired hepatic function
3. Glitazone, glinide, and sulfonylurea group: renal failure or renal impairment defined as estimated glomerular filtration rate <30 ml/min (severe renal impairment) at Visit 1, Biguanide group: renal failure or renal impairment defined as estimated glomerular filtration rate <60 ml/min (moderate renal impairment) at Visit 1
4. Treatment with anti-obesity drugs

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Actual)
Dates: Start 2010-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (43):
- Japan (43):
  - 1218.78.008 Boehringer Ingelheim Investigational Site, Akishima, Tokyo
  - 1218.78.030 Boehringer Ingelheim Investigational Site, Amagasaki, Hyogo
  - 1218.78.017 Boehringer Ingelheim Investigational Site, Annaka, Gunma
  - 1218.78.006 Boehringer Ingelheim Investigational Site, Aomori, Aomori
  - 1218.78.007 Boehringer Ingelheim Investigational Site, Aomori, Aomori
  - 1218.78.009 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1218.78.013 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1218.78.032 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 1218.78.040 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 1218.78.037 Boehringer Ingelheim Investigational Site, Higashi Osaka, Osaka
  - 1218.78.043 Boehringer Ingelheim Investigational Site, Hitachinaka, Ibaraki
  - 1218.78.019 Boehringer Ingelheim Investigational Site, Isesaki, Gunma
  - 1218.78.036 Boehringer Ingelheim Investigational Site, Kashiwara, Osaka
  - 1218.78.026 Boehringer Ingelheim Investigational Site, Kasugai, Aichi
  - 1218.78.038 Boehringer Ingelheim Investigational Site, Kawachinagano, Osaka
  - 1218.78.021 Boehringer Ingelheim Investigational Site, Kitaazumi-gun, Nagano
  - 1218.78.022 Boehringer Ingelheim Investigational Site, Matsumoto, Nagano
  - 1218.78.033 Boehringer Ingelheim Investigational Site, Matsumoto, Nagano
  - 1218.78.012 Boehringer Ingelheim Investigational Site, Meguro-ku, Tokyo
  - 1218.78.041 Boehringer Ingelheim Investigational Site, Meguro-ku, Tokyo
  - 1218.78.034 Boehringer Ingelheim Investigational Site, Morioka, Iwate
  - 1218.78.035 Boehringer Ingelheim Investigational Site, Morioka, Iwate
  - 1218.78.018 Boehringer Ingelheim Investigational Site, Moriya, Ibaraki
  - 1218.78.024 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1218.78.025 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1218.78.027 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1218.78.028 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1218.78.031 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1218.78.039 Boehringer Ingelheim Investigational Site, Oita, Oita
  - 1218.78.004 Boehringer Ingelheim Investigational Site, Okinawa, Okinawa
  - 1218.78.016 Boehringer Ingelheim Investigational Site, Sagae, Yamagata
  - 1218.78.001 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1218.78.020 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1218.78.042 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1218.78.005 Boehringer Ingelheim Investigational Site, Shimajiri-gun, Okinawa
  - 1218.78.014 Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - 1218.78.002 Boehringer Ingelheim Investigational Site, Shinjyuku-ku. Tokyo
  - 1218.78.011 Boehringer Ingelheim Investigational Site, Shizuoka, Shizuoka
  - 1218.78.003 Boehringer Ingelheim Investigational Site, Suita, Osaka
  - 1218.78.023 Boehringer Ingelheim Investigational Site, Tokorozawa, Saitama
  - 1218.78.029 Boehringer Ingelheim Investigational Site, Tokorozawa, Saitama
  - 1218.78.010 Boehringer Ingelheim Investigational Site, Tsuchiura, Ibaraki
  - 1218.78.015 Boehringer Ingelheim Investigational Site, Yamagata, Yamagata

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 618 patients were enrolled in the trial at 43 trial sites, and 37 patients were withdrawn from the trial because of screening failure. 581 patients were entered into the 2-week placebo run-in period, and 7 patients were withdrawn. 574 patients completed the 2-week placebo run-in period and took linagliptin 5 mg or metformin.
Period: Overall Study
Arm/Group | Bigu+Lina | Glin+Lina | Glit+Lina | SU+Lina | A-GI+Lina | SU+Met | A-GI+Met
Started | 82 | 66 | 74 | 143 | 85 | 63 | 61
Completed | 79 | 58 | 69 | 132 | 83 | 58 | 59
Not Completed | 3 | 8 | 5 | 11 | 2 | 5 | 2
Not completed — Adverse Event | 2 | 6 | 0 | 7 | 1 | 4 | 0
Not completed — Protocol Violation | 1 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 2 | 1 | 1 | 1 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Other (house moving) | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bigu+Lina | Glin+Lina | Glit+Lina | SU+Lina | A-GI+Lina | SU+Met | A-GI+Met | Total
Number analyzed (Participants) | 82 | 66 | 74 | 143 | 85 | 63 | 61 | 574
Age, Customized [Mean (Standard Deviation); unit: years] | 58.4 (9.9) | 62.6 (8.8) | 60.4 (9.4) | 61.8 (10.8) | 62.0 (10.4) | 61.2 (10.6) | 59.3 (10.3) | 60.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 18 | 16 | 38 | 30 | 19 | 19 | 173
  Male | 49 | 48 | 58 | 105 | 55 | 44 | 42 | 401

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs)
Description: The number of patient with any AEs, patients with severe AE, patients with AEs leading to discontinuation of trial drug, and patients with Hypoglycaemic events
Time Frame: The first drug administration through 7 days after the last drug administration, up to 382 days
Population: The treated set (TS) comprised all patients who received at least one dose of randomised study medication in the 52-week treatment period
Measure: Number; unit: Patients
Arm/Group | Bigu+Lina | Glin+Lina | Glit+Lina | SU+Lina | A-GI+Lina | SU+Met | A-GI+Met
Number analyzed (Participants) | 82 | 66 | 74 | 143 | 85 | 63 | 61
Patients
  Patients with any AE | 69 | 55 | 62 | 114 | 71 | 44 | 52
  Patients with severe AE | 1 | 1 | 0 | 2 | 1 | 1 | 0
  Patients with AEs leading to discontinuation | 2 | 5 | 0 | 8 | 1 | 4 | 0
  Patients with Hypoglycaemic events | 1 | 0 | 2 | 21 | 2 | 10 | 2

2. Secondary Outcome: Glycosylated Haemoglobin A1c (HbA1c)
Description: The change from baseline in HbA1c after 52 weeks of treatment. When the HbA1c after 52 weeks treatment was missing, the value from the measurements at the closest preceding visit replaced the missing value.
Time Frame: Baseline and 52 weeks
Population: The full analysis set (FAS) comprised all treated patients who had baseline HbA1c measurement and at least one on-treatment HbA1c measurement available
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Bigu+Lina | Glin+Lina | Glit+Lina | SU+Lina | A-GI+Lina | SU+Met | A-GI+Met
Number analyzed (Participants) | 82 | 63 | 73 | 140 | 85 | 62 | 61
Percentage
  Baseline | 7.98 (0.75) | 7.92 (0.82) | 7.86 (0.83) | 8.12 (0.78) | 7.87 (0.75) | 8.01 (0.64) | 8.07 (1.04)
  At 52 weeks | 7.10 (0.82) | 7.19 (0.75) | 7.07 (0.74) | 7.42 (0.91) | 6.96 (0.75) | 7.19 (0.72) | 6.98 (0.75)
  Change from baseline to 52 weeks | -0.88 (0.64) | -0.73 (0.65) | -0.79 (0.50) | -0.70 (0.70) | -0.91 (0.61) | -0.82 (0.78) | -1.09 (0.87)

ADVERSE EVENTS:
Time Frame: The first drug administration through 7 days after the last drug administration, up to 382 days
Arm/Group | Bigu+Lina | Glin+Lina | Glit+Lina | SU+Lina | A-GI+Lina | SU+Met | A-GI+Met
Serious Adverse Events (participants affected / at risk) | 8/82 | 5/66 | 2/74 | 7/143 | 7/85 | 5/63 | 3/61
Other Adverse Events (participants affected / at risk) | 55/82 | 41/66 | 37/74 | 83/143 | 54/85 | 31/63 | 33/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bigu+Lina (N=82) | Glin+Lina (N=66) | Glit+Lina (N=74) | SU+Lina (N=143) | A-GI+Lina (N=85) | SU+Met (N=63) | A-GI+Met (N=61)
Infectious peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lip and/or oral cavity cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bigu+Lina (N=82) | Glin+Lina (N=66) | Glit+Lina (N=74) | SU+Lina (N=143) | A-GI+Lina (N=85) | SU+Met (N=63) | A-GI+Met (N=61)
Nasopharyngitis (Infections and infestations) | 30 | 30 | 25 | 45 | 35 | 13 | 27
Bronchitis (Infections and infestations) | 9 | 1 | 1 | 5 | 3 | 1 | 3
Pharyngitis (Infections and infestations) | 5 | 5 | 3 | 5 | 2 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 2 | 1 | 0 | 2 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 2 | 4 | 4 | 4 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 20 | 1 | 10 | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 6 | 4 | 3 | 0 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 4 | 0
Constipation (Gastrointestinal disorders) | 3 | 3 | 2 | 4 | 5 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1 | 1 | 3 | 4 | 1
Contusion (Injury, poisoning and procedural complications) | 4 | 2 | 1 | 10 | 2 | 1 | 5
Fall (Injury, poisoning and procedural complications) | 4 | 3 | 1 | 10 | 3 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 4 | 1 | 3 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 1 | 1 | 0 | 8 | 3 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 4 | 5 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes